CLINICAL TRIAL: NCT02980068
Title: An Open Label Study of Oral Nitrate in Adults With Pulmonary Hypertension With Heart Failure and Preserved Ejection Fraction (PH-HFpEF) and Normal Healthy Adults
Brief Title: A Study of Oral Nitrate in Adults With Pulmonary Hypertension With Heart Failure and Preserved Ejection Fraction
Acronym: PMED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19120066; 5P01HL103455 (NIH)
Record Dates: First submitted 2016-11-17; First posted 2016-12-02 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary; Hypertension; Heart Failure; Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 15N Nitrate (Experimental): single 1,000mg dose of 15N nitrate with 3g of conjugated linoleic acid (CLA).
  Interventions: Drug: 15N Nitrate
- 14N Sodium Nitrate (Experimental): single 1,000mg dose of 14N sodium nitrate with 3g of conjugated linoleic acid (CLA)
  Interventions: Drug: 14N Nitrate

INTERVENTIONS:
Drug: 15N Nitrate — 1,000 mg/11.8 mmol, oral, on day one, hour zero
  Other Names: 15N Sodium Nitrate
  Arms: 15N Nitrate
Drug: 14N Nitrate — 1,000 mg/11.18 mmol, oral, on day hour, hour zero
  Other Names: 14N Sodium Nitrate
  Arms: 14N Sodium Nitrate

SUMMARY:
This is an open-label, single-center study to examine distinguishing features of the structure and function of the oral and gut microbiome in healthy adult normal volunteers compared to volunteers with PH-HFpEF in the breakdown of oral nitrate.

DETAILED DESCRIPTION:
We will enroll 60 Group II PH (PH-HFpEF) or Group I PAH patients and 60 matched healthy controls over three years. The Subjects will receive a single dose of one of the two study drugs, determined by whether they will participate in one study visit or two: 15N nitrate (1,000 mg) or 14N Sodium Nitrate: standard sodium nitrate, and all will receive one dose of CLA 3g. Twenty of the PH or PAH subjects and 20 of the control subjects willing to return for a follow up visit 24 hours after drug administration will receive 15N nitrate. All others will receive standard sodium nitrate. CLA will be obtained from GNC (General Nutrition Corporation) and given once.

Throughout the experiment, we will measure blood pressure, heart rate, and respiratory rate as well as co-oximetry. Plasma samples are collected at approximate times 0, 2, and 6 hrs post-drug administration. Urine will be collected at approximate times 0 and 6 hrs. We will examine plasma and urine nitrate and nitrite. The 40 subjects who return for a second visit 24 hours post-drug administration will provide an additional plasma and urine sample.

ELIGIBILITY:
INCLUSION:

* Male or female, 18 years of age or older
* PH group: Pulmonary hypertension, hemodynamically defined by a mean PAP ≥ 25 mm Hg, and a TPG >= 12 at rest or during exercise as demonstrated on a right heart catheterization in the last 10 years
* RHC Control group: Normal hemodynamics (mean PAP < 25 mm Hg, PCWP ≤ 15 mm Hg) on clinical right heart catheterization
* Healthy Control group: Healthy patients with no evidence of pulmonary hypertension, respiratory or cardiac disease
* Ability to provide written informed consent

EXCLUSION:

* Use of systemic antibiotics and/or chlorhexidine mouthwash, within the previous three months
* Use of immune suppression (chemotherapy, oral prednisone greater than 20mg per day, etc) with in the previous three months
* Use of phosphodiesterase-5 inhibitors (tadalafil, sildenafil, etc) within 7 days before study drug administration
* Current pregnancy or lactation
* Uncontrolled systemic hypertension based on repeated measurement of sitting systolic blood pressure >185 mm Hg or sitting diastolic blood pressure >110 mm Hg at screening
* Has chronic renal insufficiency as defined by serum creatinine >3 mg/dL at screening or requires dialytic support
* Known history of left ventricular ejection fraction < 40% by multiple gated acquisition scan (MUGA), angiography, or echocardiography
* History of atrial septostomy
* Repaired or unrepaired congenital heart disease
* Pericardial constriction
* Restrictive or constrictive cardiomyopathy
* Symptomatic coronary disease with demonstrable ischemia
* Addition or change in dosing of hormonal contraception medications (OCP, IUD, Depo-Provera) in the past 4 weeks.
* Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study or would prevent completion of the study
* Active participation in other research studies with investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change in nitrate level in urine | Urine collected approx 0 & 6 hours after drug administration
  The investigators will examine urine nitrate
Change in nitrate level in plasma | Approx 50cc of blood drawn approx 0, 2, & 6 hours after drug administration
  The investigators will examine plasma nitrate
Bacterial content of gut microbiome | Stool collected before drug administration
  Stool will be analyzed for bacterial makeup
Bacterial content of the oral microbiome | Saliva and tongue scraping will occur preceding administration of drug
  Saliva and tongue scraping will be analyzed for bacterial makeup
Change in nitrite level in urine | Urine collected approx 0 & 6 hours after drug administration
  The investigators will examine urine nitrite
Change in nitrite level in plasma | Approx 50cc of blood drawn approx 0, 2, & 6 hours after drug administration
  The investigators will examine plasma nitrite

SECONDARY OUTCOMES:
Change in blood pressure | Frequently over 6 hour study visit
Change in heart rate | Continuous over 6 hour study visit
Change in respiratory rate | Continuous over 6 hour study visit
Change in hemoglobin concentration | Continuous over 6 hour study visit

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nydia Chien, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
After de-identification, all participant data collected during the trial will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made following publication.
Access Criteria: Data will be available publicly.